CLINICAL TRIAL: NCT03410602
Title: Effect on Nonsurgical Periodontal Therapy on First Molars Banded for Fixed Orthodontic Treatment
Brief Title: Nonsurgical Periodontal Therapy on Banded First Molars
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MADC/IRB-IX/2016/153
Record Dates: First submitted 2018-01-04; First posted 2018-01-25 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Periodontitis
Keywords: Nonsurgical periodontal therapy; Orthodontic bands
MeSH Terms: conditions — Periodontitis | interventions — Dental Scaling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supragingival and subgingival scaling (Placebo Comparator): Supragingival and subgingival scaling group comprised of 15 orthodontic patients treated with routine full-mouth supragingival scaling and subgingival scaling only around all banded first molars. Parameters such as radiographic evidence of alveolar crestal bone level, gingival index, probing pocket depth and clinical attachment level around the banded first molars and full-mouth plaque index were recorded as a change from baseline to 12th month.
  Interventions: Procedure: Full-mouth supragingival scaling; Procedure: Subgingival scaling
- Subgingival irrigation (Active Comparator): Subgingival irrigation group comprised of 15 orthodontic patients treated with full-mouth supragingival scaling and subgingival scaling only around all banded first molars followed by irrigation with 0.2% chlorhexidine gluconate solution (Trade name: HEXIDINE), an antiseptic - antiplaque agent. Parameters such as radiographic evidence of alveolar crestal bone level, gingival index, probing pocket depth and clinical attachment level around the banded first molars and full-mouth plaque index were recorded as a change from baseline to 12th month.
  Interventions: Procedure: Full-mouth supragingival scaling; Procedure: Subgingival scaling; Drug: Subgingival irrigation

INTERVENTIONS:
Procedure: Full-mouth supragingival scaling — Control group comprised of 15 patients who were treated with routine full-mouth supragingival scaling.
  Other Names: Oral prophylaxis
Procedure: Subgingival scaling — Test group comprised of 15 patients who were treated with subgingival scaling only around all banded first molars.
  Other Names: Deep scaling
Drug: Subgingival irrigation — Test group comprised of 15 patients who were treated with subgingival irrigation only around all banded first molars with 0.2% chlorhexidine gluconate solution (Trade name: HEXIDINE), an antiseptic - antiplaque agent.
  Other Names: Chemical plaque control
  Arms: Subgingival irrigation

SUMMARY:
The aim of this study was to evaluate the effect of nonsurgical periodontal therapy on first molars banded for fixed orthodontic treatment.

DETAILED DESCRIPTION:
A total of 30 patients who were about to undergo fixed orthodontic therapy were selected and divided into two groups.

Group A comprised of 15 patients who were treated with routine full-mouth supragingival scaling and subgingival scaling only around all banded first molars.

Group B comprised of 15 patients who were treated with full-mouth supragingival scaling and subgingival scaling only around all banded first molars followed by irrigation with 0.2% chlorhexidine gluconate solution (Trade name: HEXIDINE), an antiseptic - antiplaque agent. Treatment for both the groups was performed at 3rd month, 6th month and 9th month.

Parameters such as radiographic evidence of alveolar crestal bone level, gingival index, probing pocket depth and clinical attachment level around the banded first molars and full-mouth plaque index were recorded as a change from baseline to 12th month. The differences between the values were assessed and sent for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients within the age group 16 to 25 years.
2. Patients diagnosed with malocclusion undergoing fixed orthodontic treatment having banded first molars.
3. Systemically healthy patients.

Exclusion Criteria:

1. Congenital malformations in the oral cavity.
2. Patients who had undergone periodontal therapy within the previous 6 months.
3. Patients using removable orthodontic appliances.
4. Patients who were administered antibiotics or other systemic or topical antimicrobial agents.
5. Smokers.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline radiographic evidence of alveolar crestal bone level at 12th month | Baseline to 12th month
  Radiographic evidence of alveolar crestal bone level was measured around each banded first molar

SECONDARY OUTCOMES:
Change from baseline plaque index at 12th month | Baseline to 12 month
  Full-mouth plaque index measurements were carried out at four sites around each tooth (mesiobuccal, buccal, distobuccal and lingual).
Change from baseline gingival index at 12th month | Baseline to 12th month
  The measurements were carried out around all the banded first molars at four sites (mesiobuccal, buccal, distobuccal and lingual).
Change from baseline probing pocket depth at 12th month | Baseline to 12th month
  The probing pocket depth was measured clinically using Williams periodontal probe at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, distolingual and lingual) of each banded first molar.
Change from baseline clinical attachment level at 12th month | Baseline to 12th month
  Clinical attachment level (CAL) was measured as the distance between a fixed point on the crown such as cementoenamel junction to the base of the pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Nashra Kareem, BDS, Principal Investigator — Meenakshi Ammal Dental College and Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babay N, Al Jasser N. Subgingival irrigation effects of chlorhexidine or sanguinarine on gingivitis in orthodontic patients. J Clin Pediatr Dent. 1996 Spring;20(3):225-8. PMID 8634210
- [Background] Morrow D, Wood DP, Speechley M. Clinical effect of subgingival chlorhexidine irrigation on gingivitis in adolescent orthodontic patients. Am J Orthod Dentofacial Orthop. 1992 May;101(5):408-13. doi: 10.1016/0889-5406(92)70113-O. PMID 1590289